CLINICAL TRIAL: NCT05752279
Title: Balanced Multi-electrolyte Solution Versus 0.9% Sodium Chloride as Fluid Therapy for Patients Presenting With Moderate to Severe Diabetic Ketoacidosis
Brief Title: Balanced Multi-Electrolyte Solution Versus Saline Trial for Diabetic KetoAcidosis
Acronym: BEST-DKA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The George Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TGI CCP-2378-352
Record Dates: First submitted 2023-02-07; First posted 2023-03-02 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Ketoacidosis
MeSH Terms: conditions — Diabetic Ketoacidosis | interventions — Plasma-lyte 148; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plasma-Lyte® 148 (Active Comparator): Plasma-Lyte® 148 fluid 1L given intravenously for fluid replacement
  Interventions: Drug: Plasma-Lyte 148
- 0.9% sodium chloride (Active Comparator): Normal saline fluid 1L given intravenously for fluid replacement
  Interventions: Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: Plasma-Lyte 148 — Plasma-Lyte® 148 intravenous fluid for resuscitation in patients with keto-acidosis
  Other Names: Balanced multi-electrolyte solution
  Arms: Plasma-Lyte® 148
Drug: 0.9% sodium chloride — 0.9% sodium chloride intravenous fluid for resuscitation in patients with keto-acidosis
  Other Names: normal saline
  Arms: 0.9% sodium chloride

SUMMARY:
The goal of this blinded, cluster cross-over, randomised controlled trial is to determine whether fluid therapy with Plasma-Lyte® 148 increases the number of days alive and days out of hospital to day-28 compared to 0.9% sodium chloride ('0.9% saline') in critically ill patients presenting to the Emergency Department (ED) and deemed to require admission to a critical care area (ICU, HDU) with moderate to severe diabetic ketoacidosis (DKA).

DETAILED DESCRIPTION:
DKA is a life-threatening complication of diabetes mellitus, described in patients with both type-1 diabetes, and type-2 diabetes(1). Data from the Australian Institute of Health and Welfare suggest that between 2009-10 to 2014-15, there has been a 21% increase in the hospitalisation amongst young people with DKA(2). An interrogation of the Australian and New Zealand Intensive Care Society (ANZICS) Centre for Outcomes Research (CORE) database revealed that the incidence of ICU admission of patients with DKA in Australia and New Zealand increased 5-fold between 2000 and 2013 (0.97/100000, 95%CI 0.84 to1.10) in 2000 to (5.3/100000, 95%CI 4.98to 5.53, (P<0.0001)(3).

Increasing incidences were observed predominantly in rural and metropolitan hospitals (Figure 1), about 88% of the admissions to the ICU were from the ED. The median (IQR) ICU and hospital length of stay were 1.8 (1-2.8) and 4 (2.6-7.4) days respectively. Recent data from the ANZICS-CORE database confirmed the persistent high admission rate of severe DKA to Australian ICUs - 2849 and 2862 admissions in 2019 and 2020.

A major review of DKA management protocols in 2017 concluded that there are major deficiencies in evidence for optimal management of DKA(33). Current practice is guided by weak evidence and consensus opinion.

Studies comparing Plasma-Lyte® 148 vs. 0.9% saline in DKA demonstrate a trend towards a more rapid resolution of acidosis, equivalent glucose control and stable ketones with Plasma-Lyte® 148. In addition, there are trends towards reduced length of ICU and hospital stay with the use of Plasma-Lyte® 148.

Given the clinical uncertainty and substantial variability in practice. there is a scientific, clinical and health economic imperative to conduct a high-fidelity study to provide definitive evidence to inform clinicians regarding the choice of resuscitation fluids for patients with DKA. BEST-DKA will address this critical knowledge gap.

BEST-DKA is a multi-centre, blinded, cluster-crossover trial conducted in 20 Australian hospitals, consisting of two 12-month intervention periods with a one-month inter-period gap.

Each hospital is a single cluster, with all patients admitted with DKA to that hospital's ED during the intervention periods will potentially be eligible for inclusion in the trial. After the first 12-month intervention period during which recruited patients will receive either Plasma-Lyte® 148 or 0.9% saline, there will be a one-month inter-period gap during which patients will not be recruited into the trial. Following this each critical care area will change to using the fluid to which they were not assigned for the first period (Figure 4). All included patients will receive blinded fluids (Plasma-Lyte® 148 or 0.9% saline) as part of their DKA therapy depending on the fluid assigned to the site for the relevant intervention period.

Both study fluids are manufactured by Baxter Healthcare Pty Ltd (Old Toongabbie, NSW) and will be labelled, packed and distributed by the company directly to the study sites in periodic shipments. Study fluid will be coded and labelled in compliance with applicable regulations, and in a manner that protects the blinding.

All clinicians involved in the prescription of blinded study treatment must read Product Information for both Plasma-Lyte® 148 and 0.9% saline which provide detailed information about the composition, indications, side effects, suggested dosage and contraindications of the study treatments.

The volume and rate of blinded study fluid administered will be guided by the standard clinical endpoints determined by the treating clinician. Study treatments will be started following study enrolment and continue until discharge from a critical care area or for a maximum of 72 hrs, whichever is earlier. If patients are re-admitted to the critical care area within 72 hours with a relapse of ketoacidosis, the clinician may use open label fluids for the managements of ketoacidosis. within 72 hours they will continue to receive blinded treatment fluid. Glucose containing solutions can be added in as required for blood glucose or ketosis management. The use of bicarbonate therapy and the need for potassium, phosphate and magnesium supplementation will be at the discretion of the treating clinician and data on its use will be collected.

The primary outcome will be evaluated at day-28 and patients contacted via telephone.

End-user/consumer representatives have been involved in all components of the research program including protocol development, choice of primary outcome, funding applications, and membership of the management committee. End-user/consumer representatives will continue to be involved in the conduct of the study and play a key role in the dissemination of results. Currently, membership of the study management committee includes the President of the advocacy group, Diabetes Australia; Director of Australian Centre for Accelerating Diabetes Innovations (ACADI); and a consumer who lives with diabetes.

This study aligns with the Medical Research Future Fund (Australia Government grant) funded ACADI objective to address the acute complications of diabetes including management of DKA.

The study has been endorsed by the Australasian College for Emergency Medicine (ACEM) and a letter of support from for the study from Diabetes Australia.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the ED with a primary diagnosis of moderate to severe DKA for whom both saline and Plasma-Lyte® 148 are considered appropriate fluids
* Blood glucose level > 14mmol/L
* pH < 7.25
* Serum bicarbonate <15 mmol/L
* Elevated anion gap > 12mEq/L
* Ketones positive on finger prick measurements
* In the judgement of the treating clinician critical care area admission is required

Exclusion Criteria:

* Age less than 18 years
* Patients who have received more than 2000ml of non study fluid prior to study enrolment
* Serum Na > 155 or <120 mmol/L
* Contraindication to either study fluid e.g. previous allergic reaction to Plasma-Lyte® 148
* Patients with hyperosmotic hyperglycaemic non-ketotic syndrome
* Other clinical conditions that preclude large volumes of fluid resuscitation
* Previous inclusion in BEST-DKA trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Hospital free days (HFD) up to day-28 after study enrolment | from time of enrolment to 28 days
  Number of hospital free days from time of hospital discharge

SECONDARY OUTCOMES:
ICU free days up to 28 days after study enrolment | 28 days after enrolment
  Number of ICU free days from time of ICU discharge
ICU and hospital readmissions up to 28 days after study enrolment | 28 days after enrolment
  Number of days free from ICU and hospital from time of hospital discharge
Acute kidney injury assessed by comparing serum creatinine using Kidney Disease: Improving Global Outcomes (KDIGO) criteria | 28 days after enrolment
  injury assessed by comparing change in serum creatinine using Kidney Disease: Improving Global Outcomes (KDIGO) criteria
Episodes of post-study enrolment decrease in Glasgow Coma Scale (GCS) by more than 2 in the first 24 hours | first 24 hours from enrolment
  decrease in Glasgow Coma Score by more than 2 points
Time to resolution of ketosis | from time of enrolment to day 28
  resolution of acidosis
Cumulative insulin dosage in the first 48 hours | first 48 hours from time of enrolment
  Total amount of insulin given to the patient from enrolment to 48 hours
Duration of IV insulin infusion | from time of enrolment to day 28
  Total amount of IV insulin given to the patient from time of enrolment to day 28
Cumulative potassium replacement | from time of enrolment to day 28
  Total amount of potassium given to the patient from time of enrolment to day 28

OTHER OUTCOMES:
Cost-effectiveness | from time of enrolment to day 28
  Calculation of the incremental cost-effectiveness ratios

CONTACTS AND LOCATIONS:
Locations (21):
- Australia (21):
  - Blacktown Hospital, Blacktown, New South Wales
  - Camperdown Hospital, Camperdown, New South Wales
  - Dubbo Base Hospital, Dubbo, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Maitland Hospital, Metford, New South Wales
  - Orange Hospital, Orange, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Caboolture Hospital, Caboolture, Queensland
  - Queen Elizabeth II Jubilee Hospital, Coopers Plains, Queensland
  - Redcliffe Hospital, Redcliffe, Queensland
  - Rockhampton Hospital, Rockhampton, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Ballarat Base Hospital, Ballarat, Victoria
  - Monash Health-Casey Hospital, Berwick, Victoria
  - Dandenong Hospital, Dandenong, Victoria
  - Frankston Hospital - Peninsula Health, Frankston, Victoria
  - Latrobe Regional Hospital, Traralgon, Victoria

IPD SHARING:
Plan to Share IPD: Undecided